CLINICAL TRIAL: NCT00788853
Title: DiabCare Asia 2008. A Cross-sectional Survey to Evaluate Diabetes Management, Control, Complications, Psychosocial Aspects of Diabetic Patients in Asia and to Evaluate Perceptions and Practices of Physicians and Patients About Diabetes Management in Asia. DiabCare Asia 2008 - Indonesia
Brief Title: A Survey to Evaluate Diabetes Management, Control, Chronic Complications, Psychosocial Aspects of Diabetic Subjects in Indonesia
Acronym: DiabCare Asia
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: INS-3677
Record Dates: First submitted 2008-11-10; First posted 2008-11-11 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
Keywords: DiabCare Asia 2008, Cross-sectional survey, Glycemic control, Psychosocial well-being, Diabetic complications, Quality of life.
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Complications

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — No treatment is given

SUMMARY:
This study is conducted in Asia. The aim of this observational study is to evaluate current status of diabetes management, control, complications in diabetic subjects in Asia. Further perceptions and practices of physicians and subjects about diabetes management in Asia will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients registered in the particular centre for more than 12 months.
* Patients should have visited the centre at least once in the last 3-6 months before the initial study visit.
* Patients willing to sign informed consent form.

Exclusion Criteria:

* Repetition of any patient as patients should not be included twice for any reason.
* Unwilling to participate or unable to comply with protocol requirements.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with diabetes mellitus (both type 1 and type 2) being treated at general hospitals, diabetes clinics and referral clinics will be selected according to inclusion and exclusion criteria. Patients will be selected randomly from clinic record/list to avoid any bias.
Sampling Method: Non-Probability Sample
Enrollment: 1832 (Actual)
Dates: Start 2008-11; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Mean age of onset of either type 1 or type 2 diabetes mellitus | study visit
Mean duration of treatment of type 2 diabetes mellitus. | study visit
Percentage of patients on either insulin therapy or OAD (oral anti-diabetic drug) therapy. | study visit
Mean duration of diabetes in type 1 and type 2 diabetes patients respectively. | study visit
Mean FPG (fasting plasma glucose),PPG (post prandial glucose) and HbA1c of diabetic patients. | study visit
Percentage of diabetic patients with HbA1c target below or equal to 7.0%. | study visit
Percentage of diabetic patients with HbA1c target below or equal to 6.5%. | study visit
Percentage of diabetic patients having dyslipidemia and hypertension | study visit
Percentage of diabetic patients having cardiovascular complications | study visit
Percentage of diabetic patients having peripheral vascular disease | study visit
Percentage of diabetic patients having diabetic nephropathy | study visit
Percentage of diabetic patients having diabetic eye complications | study visit

SECONDARY OUTCOMES:
Patients' perception will be analysed through Patient questionnaire measuring:Psychological well-being, Quality of life and Patients' compliant to treatment | study visit
Physician questionnaire measuring awareness about:HbA1c test and its goal, Anti-diabetic treatment and Barriers towards optimum diabetes control | study visit
Duration of diabetes associated with highest number of diabetic complications | study visit
Minimum duration of diabetes associated with 10% incidence of diabetic complications (CVD, nephropathy and retinopathy) | study visit

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Jakarta, Indonesia

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com